CLINICAL TRIAL: NCT02867176
Title: Pain Management in Corneal Collagen Crosslinking for Keratoconus: Prospective Randomized Study
Brief Title: Pain Management in Corneal Collagen Crosslinking for Keratoconus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CXL-PAIN
Record Dates: First submitted 2016-08-03; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Gabapentin; Ketorolac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corneal collagen CXL epi-off (Other): For the epithelium-off procedure, the corneal epithelium is removed with a 10-minute soak time with isotonic riboflavin 0.1% solution and 4 minutes of exposure with 30 mw/cm2 ultraviolet-A irradiation.
  Interventions: Drug: Gabapentin; Drug: Ketorolac
- Corneal collagen CXL epi-on (Other): For the epithelium-on procedure, riboflavin is applied for a total soak of 4 minutes; the cornea is then completely rinsed with additional riboflavin for a total of 6 minutes. The ultraviolet-A irradiation is performed for 2 minutes and 40 seconds at 45mw/cm2.
  Interventions: Drug: Gabapentin; Drug: Ketorolac

INTERVENTIONS:
Drug: Gabapentin — The gabapentin (Neurontin, Pfizer, Mexico) group was instructed to take one 300-mg capsule the night before surgery and 1 capsule every 8 hours on the day of surgery and for the first 3 postoperative days.
  Other Names: Neurontin
Drug: Ketorolac — The ketorolac group (Dolac, Siegfried Rhein, Mexico) was instructed to take their 10-mg tablets every 8 hours on the day of surgery and for the first 3 postoperative days.
  Other Names: Dolac

SUMMARY:
This is a prospective, randomized, single blind study. Patients enrolled in the study were randomly assigned to a ketorolac or a gabapentin group for pain control. Different pain scores and variables will be evaluated, along with others side effects variables.

DETAILED DESCRIPTION:
This is a prospective, randomized, single blind study. Patients enrolled in the study were randomly assigned to the ketorolac or gabapentin group. The gabapentin (Neurontin, Pfizer, Mexico) group was instructed to take one 300-mg capsule the night before surgery and 1 capsule every 8 hours on the day of surgery and for the first 3 postoperative days. The ketorolac group (Dolac, Siegfried Rhein, Mexico) was instructed to take their 10-mg tablets every 8 hours on the day of surgery and for the first 3 postoperative days. Different pain scores and variables will be evaluated, along with others side effects variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with keratoconus older than 18 years with documented bilateral keratometric progression in the previous 6 to 12 months.

Exclusion Criteria:

* Previous ocular or systemic diseases that could affect epithelial healing; use of topical or systemic non-steroidal anti-inflammatory drugs, or chronic use of any other pain medication, pregnancy and allergy to the drugs of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Numeric scale of pain | 5 days
  Using a numeric scale of pain, patients were asked to state their pain intensity on a scale of 0 to 10, explaining the patient that a 0 represents no pain at all and a 10 would be the worst pain imaginable.

SECONDARY OUTCOMES:
Side effects | 5 days
  The last four issues on the questionnaire were related to side effects associated with the use of the medication, specifically dizziness, drowsiness, headaches, and gastrointestinal symptoms
Symptoms related to pain | 5 days
  Patients were asked to rate the severity of four different symptoms during the 24-hour period prior to follow-up: tearing, light sensitivity, foreign body sensation, and discomfort/irritation

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Graue-Hernandez, Md, MSc, Study Chair — Instituto de Oftalmologia Conde de Valenciana

IPD SHARING:
Plan to Share IPD: No